CLINICAL TRIAL: NCT05521152
Title: Prophylactic Use of Norepinephrine for Prevention of Intraoperative Hypotension in Infants Undergoing Kasai Portoenterostomy Operation for Biliary Atresia: Double Blinded Randomized Controlled Trial
Brief Title: Norepinephrine for Prevention of Intraoperative Hypotension in Infants Undergoing Kasai Portoenterostomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator,Lecturer of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-12-2021
Record Dates: First submitted 2022-08-28; First posted 2022-08-30 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia; Pediatrics; Biliary Atresia
Keywords: Kasai; biliary atresia; norepinephrine; hypotension
MeSH Terms: conditions — Biliary Atresia; Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group N) (Experimental): 1 mg norepinephrine will be diluted in dextrose 5% in a 50 mL syringe using a nomogram based on the infant body weight so that 1mL= 0.05 µg/kg/min norepinephrine infusion and the syringe will be set on 2 ml/h
  Interventions: Drug: Norepinephrine Bitartrate
- (Group S) (Placebo Comparator): equivalent volume of saline will be prepared in 50 mL syringe and the infusion will be set on 2ml/kg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norepinephrine Bitartrate — anesthesia resident (who will not be involved in patient management to ensure the blinding) will be responsible for preparing norepinephrine infusion or placebo as instructed in the envelope as follow: 1 mg norepinephrine will be diluted in dextrose 5% in a 50 mL syringe using a nomogram based on the infant body weight so that 1mL= 0.05 µg/kg/min norepinephrine infusion.
  the attending anesthetist will be instructed to set the 2 syringe pumps on 2 mL/h continuous infusion following skin incision.
  Arms: (Group N)
Drug: Placebo — Placebo
  Arms: (Group S)

SUMMARY:
This study aims to assess the efficacy and safety of prophylactic intraoperative norepinephrine infusion versus the standard technique on decreasing the incidence of intraoperative hypotension in infants undergoing Kasai portoenterostomy operation.

DETAILED DESCRIPTION:
All children will be anesthetized in accordance with the local policy of pediatric anesthesia unit in Abu El-Reesh pediatric hospital-Cairo university.

Upon arrival to the operating room heart rate HR, noninvasive blood pressure NBP and oxygen saturation SPO2 will be monitored using standard monitor (Dräger infinity vista XL) before inhalational induction of anesthesia using titration of sevoflurane in oxygen air mixture 60% (starting from 3% up to 8%) until the child is put to sleep.

After securing an intravenous line anesthesia will be completed with 2µg/kg of fentanyl and atracurium 0.5 mg/kg to facilitate endotracheal intubation. Anesthesia will be maintained by using 1.2 % isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes. Mechanical ventilation will be set to volume-controlled mode TV:8ml/kg, I/E ratio:1/2, PEEP: 3 cmH2o and respiratory rate will be adjusted to maintain ETCO2 30-35 mmHg. Nasopharyngeal temperature probe will be inserted for monitoring of core body temperature. 22 G arterial cannula will be placed in the radial artery for continuous monitoring of arterial blood pressure and management of intraoperative hemodynamics.

Central venous catheter will be inserted under complete aseptic condition using ultrasound guidance and a Foley's catheter will be inserted in the urinary bladder.

The concealed envelopes will then be opened by an anesthesia resident (who will not be involved in patient management to ensure the blinding) and he will be responsible for preparing norepinephrine infusion or placebo as instructed in the envelope as follow:

(Group N): 1 mg norepinephrine will be diluted in dextrose 5% in a 50 mL syringe using a nomogram based on the infant body weight so that 1mL= 0.05 µg/kg/min norepinephrine infusion.

(Group S): equivalent volume of saline will be prepared in 50 mL syringe. In both groups the attending anesthetist will be instructed to set the 2 syringe pumps on 2 mL/h continuous infusion following skin incision.

Intraoperative fluid management:

All children will receive a loading dose of 10 ml/kg of lactated ringer solution over 10 minutes after induction of anesthesia and will be maintained on 10 ml/kg/h lactated ringer solution using an infusion pump. Dextrose 1% will be transfused in a separate line and rate will be adjusted according to blood glucose level.

Packed RBCs will be transfused at a dose of 15mL/kg if intraoperative Hb dropped to 8 gm/dL.

Intraoperative hemodynamic management:

Episodes of hypotension defined as reduction of the mean ABP ≥20% of the baseline mean ABP recorded preoperatively will be managed by boluses of lactated ringer solution of 10 mL/kg that will be repeated up to 30 mL/kg, if hypotension persisted, norepinephrine bolus of 0.01 µg/kg bolus will be given, if hypotension persisted after 2 boluses the surgery will be stopped and the liver will be released into the abdominal cavity until the BP is restored. Total dose of norepinephrine will be recorded.

Hypertension defined as increase of mean ABP ≥20% of the baseline mean arterial pressure ABP will be treated by stopping the infusion pump until ABP return to baseline and then the infusion will be resumed to 1 mL/h. Bradycardia defined as HR less than 80 beat/min will be managed by atropine 0.01mg/kg.

Following release of the liver the norepinephrine infusion will be stopped gradually guided by the mean ABP.

At the end of the procedure an open transverses abdominis plane block TAPB will be given using 5 mL bupivacaine 0.25% before skin closure, inhalational anesthesia will be discontinued, infusion will be stopped and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered IV after return of patient's spontaneous breathing and patients will then be transferred to PICU.

ELIGIBILITY:
Inclusion Criteria:

* Infants, ASA III, diagnosed as biliary atresia undergoing Kasai operation.

Exclusion Criteria:

* Parents refusal. Patients with complex cardiac anomalies. Patients requiring emergency or laparoscopic procedures.

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | 4 hours
  Incidence of intraoperative hypotension defined as persistent reduction of mean ABP ≥20% of the baseline mean ABP recorder preoperatively requiring release of the liver after initial resuscitation.

SECONDARY OUTCOMES:
mean arterial pressure (MAP) | 4 hours
  mean arterial pressure (MAP) will be measured upon arrival to the operating room suite as baseline and every 5 minutes after induction of anesthesia and every 3 minutes during liver mobilization till the end of surgery.
heart rate | 4 hours
  will be measured upon arrival to the operating room suite as baseline and every 5 minutes after induction of anesthesia and every 3 minutes during liver mobilization till the end of surgery.
Incidence of severe hypotension | 4 hours
  Incidence of severe hypotension defined as reduction of mean ABP ≥30% of the baseline mean ABP recorder preoperatively.
Incidence of hypertension | 4 hours
  Incidence of hypertension defined as increase of mean ABP ≥20% of the baseline
Total dose of rescue norepinephrine. | 4 hours
  Total dose of rescue norepinephrine.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarhan K, Ashraf N, Hasanin A, Zayed M, Saleh R, Elgohary M, Alkonaiesy R, Nawwar K. Norepinephrine infusion for preventing hypotension during hepatic exteriorization in Kasai portoenterostomy in infants with biliary atresia: A randomized controlled trial. Anaesth Crit Care Pain Med. 2025 May;44(3):101519. doi: 10.1016/j.accpm.2025.101519. Epub 2025 Apr 16. PMID 40250622